CLINICAL TRIAL: NCT03313973
Title: Impact of Myotensives Techniques, With and Without Auto-reeducation, on the Vital Capacity Forced by the Patient Affected by a Honeymoon Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CVF Parkinson
Record Dates: First submitted 2017-10-10; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with self stretching same muscle (Experimental)
  Interventions: Procedure: with self stretching same muscle
- with self stretching forearm muscle (Sham Comparator)
  Interventions: Procedure: with self stretching of forearm muscles

INTERVENTIONS:
Procedure: with self stretching same muscle — with self stretching
  Arms: with self stretching same muscle
Procedure: with self stretching of forearm muscles — without self stretching
  Arms: with self stretching forearm muscle

SUMMARY:
Lower respiratory tract infections are one of the main hospitalization or mortality cause in idiopathic Parkinson's disease. Because of akinesia and articular rigidity these patient develop restrictive syndrome by reduction in the thoraco-lung compliance.The consequence is a progressive loss of the aerobic physical abilities and infection.

The myotensive technique of active muscular stretching seem to increase the range of motion in healthy subject but also in patient with chronic bronchiotisis . These technics also increase the vital respiratory capacity and re enforce the muscles.So adding these technics during the period when the Parkinson's disease patient is stable would be a way of improvement .

DETAILED DESCRIPTION:
To validate if these techniques really improve the the vital respiratory capacity, investigators randomize patient in 2 groups; one will have the standard protocol of stretching + self stretching of the same muscles (experimental group) and the other one (control group) will have the standard protocol and self stretching of forearm . Self stretching of forearm is selected to avoid bias .

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* with Parkinson's disease
* stable stade of pathology
* without any treatment modification.

Exclusion Criteria:

* rehabilitation support or osteopathic support
* active smoking
* respiratory disease
* cognitives trouble
* any other neurologic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage vital respiratory capacity | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France